CLINICAL TRIAL: NCT01414465
Title: Orlistat Induced Modulation on the Fatty Acid Composition of the Red Blood Cell Membrane and Plasma Phospholipids, Triglyceride and Cholesteryl Esters in Obese Females
Brief Title: Orlistat Induced Modulation on the Fatty Acid Composition in Obese Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Germed Pharma (Industry)
Responsible Party: Bruno Geloneze, University of Campinas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIMED0010
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Overweight
Keywords: Fatty acids; orlistat; lipase; BMC (Body Mass Index) between 30 to 40 kg/m2; Women; 18 to 45 years; Premenopausal stage
MeSH Terms: conditions — Overweight | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- low caloric diet (No Intervention): 10 health obese women (BMI 30 to 40 kg/m2)
  Interventions: Drug: Orlistat
- Orlistat (Experimental): 10 obese women treated with Orlistat 120mg 3 times per day
  Interventions: Drug: Orlistat
- lifestyle counseling (Sham Comparator): Women with BMI < 30 kg/m2, no taking drug in study
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — Obese women were treated with orlistat 120mg 3 times a day for 4 months, compared with basal data and with normal weight women that didn´t receive orlistat

SUMMARY:
Orlistat is a popular drug approved for long-term use which produces weight loss by inhibiting triglycerides, main components of fats in the diet and reducing dietary fat absorption by up to 30%. The effect of this drug on human blood fatty acid profile has not been described yet. The FA composition of RBCs, plasma and platelets can be used to monitor of many pathological processes. This study presents alteration of FA composition in RBCM and phospholipids, triglycerides and cholesteryl esters from plasma of health obese female volunteers treated with nutritional orientation and orlistat (120 mg t.i.d) for 3 months.

DETAILED DESCRIPTION:
Obesity treatment requires lifestyle changes such as diet, exercise, and behavioral therapy. Orlistat is a popular drug approved for long-term use which produces weight loss by inhibiting triglycerides, main components of fats in the diet, from binding to the lipase enzyme active sites thus halting their subsequent breakdown into monoglycerides and free fatty acids necessary for fat digestion, reducing dietary fat absorption by up to 30%. The effect of this drug on human blood fatty acid profile has not been described yet.

The FA profile is typical of each lipid and tissue, however, alterations in diets, pathological processes, drugs intervention, cigarettes and alcohol consumption can alter the FA profile. The FA composition of RBCs, plasma and platelets can be used to monitor these processes. This study presents alteration of FA composition in RBCM and phospholipids, triglycerides and cholesteryl esters from plasma of health obese female volunteers treated with nutritional orientation and orlistat (120 mg t.i.d) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Obesity BMC (Body Mass Index) between 30 to 40 kg/m2 Women 18 to 45 years Premenopausal stage

Exclusion Criteria:

* Relevant diseases (diabetes, cardiovascular, gastrointestinal, renal and hepatic diseases, endocrine disorders, hemoglobinopatHy or neoplasm in the last three years)
* Chemical or natural laxatives
* Weight variation greater than 5% in the preceding 3 months
* Surgery for weight reduction
* Drugs to obesity control and/or oral corticosteroids anti-inflammatory in the last three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Orlistat induced modulation on the Fatty Acid composition in Obese Females | baseline
  This study aims to present alteration of FA composition in RBCM and phospholipids, triglycerides and cholesteryl esters from plasma of health obese female volunteers treated with nutritional orientation and orlistat (120 mg t.i.d) for 3 months.

SECONDARY OUTCOMES:
Orlistat induced modulation on the Fatty Acid composition in Obese Females | after 120 days Orlistat treatment
  This study aims to present alteration of FA composition in RBCM and phospholipids, triglycerides and cholesteryl esters from plasma of health obese female volunteers treated with nutritional orientation and orlistat (120 mg t.i.d) for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, Dr, Principal Investigator — University of Campinas (UNICAMP); Sabrina Nagassaki, Dr, Study Chair — University of Campinas (UNICAMP); Anita J Marsaioli, Dr, Study Chair — University of Campinas (UNICAMP); Thiago Inacio B Lopes, Study Chair — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/University of Campinas (UNICAMP), Campinas, São Paulo, Brazil